CLINICAL TRIAL: NCT02033577
Title: Effects of Long Biliopancreatic Limb vs Long Alimentary Limb in Superobesity
Brief Title: Effects of Long Biliopancreatic Limb Versus Long Alimentary Limb in Superobesity, a Randomized Study
Acronym: BMI>50
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aleris Obesity (Industry)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Jan Hedenbro, Senior scientist, Aleris Obesity
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCT01514799
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Severe Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Distal gastrojejunal bypass (Experimental): RYGB with 200 cm BP limb and 150 cm common limb
  Interventions: Procedure: Distal gastrojejunal bypass
- RYGB (Active Comparator): RYGB with 60 cm BP limb and 150 cm alimentary limb
  Interventions: Procedure: RYGB

INTERVENTIONS:
Procedure: Distal gastrojejunal bypass — RYGB with 200 cm BP limb and 150 cm common limb, effect on EWL, QoL and complications
  Arms: Distal gastrojejunal bypass
Procedure: RYGB — RYGB with 60 cm BP limb and 150 cm alimentary limb, effect on
  Arms: RYGB

SUMMARY:
Surgical bypassing of a longer section of the small bowel (when doing a gastric bypass operation) gives better results on body weight in the superobese. We do not yet know whether it is beneficial to exclude more of the proximal small bowel or more of the distal. Side effects of bypassing can also be different.

Study aims at clarifying possible differences in effects and side-effects of these two surgical-technical variations.

DETAILED DESCRIPTION:
Randomisation in the OR between long biliopancreatic limb and long alimentary limb. GAstric component identical.

Perioperative biopsies to assess mucosal properties at the gastrojejunostomy and the enteroanastomosis. Repeat biopsies (gastroscopy) at one year to identify changes in the mucosa at the Gastroenteroanastomosis.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 50

Exclusion Criteria:

* Psychiatric disease
* Inflammatory bowel disease
* inability to understand Swedish

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Body weight reduction | 2 years from end of inclusion
  Body weight reduction is currently the best substitute endpoint to correlate with the hard endpopints such as death, comorbidities etc.

SECONDARY OUTCOMES:
Patient assessed quality of life | 2 years from end of inclusion
  We employ SF-36, Op-9, GSRS, TFEQ scales

OTHER OUTCOMES:
Short-term complications | 0-30 days postoperatively
  Time to discharge, leaks, bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Aleris Obesity, Lund, Sweden